CLINICAL TRIAL: NCT01105936
Title: A Randomised, Double-blind, Evaluation of the Effects of Paracetamol on the BOLD fMRI Response to Painful Stimuli in Subjects With Osteoarthritis
Brief Title: Assess the Blood-Oxygen-Level-Dependent (BOLD) Signal Changes in the Brain by Paracetamol as Measured by Functional Magnetic Resonance Imaging (fMRI) in Subjects With Osteoarthritis (OA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: A3360529
Record Dates: First submitted 2010-03-04; First posted 2010-04-19 (Estimated); Results first posted 2015-03-24 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; pain; paracetamol; Blood-Oxygen-Level-Dependent functional magnetic resonance imaging
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol caplets (Experimental): Two 665 mg sustained release paracetamol caplets administered orally with water.
  Interventions: Drug: Paracetamol
- Placebo caplets (Placebo Comparator): Two placebo caplets administered orally with water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol — 665 mg sustained release paracetamol caplets
  Arms: Paracetamol caplets
Drug: Placebo — Placebo caplets
  Arms: Placebo caplets

SUMMARY:
Blood-Oxygen-Level-Dependent (BOLD) responses to painful mechanical stimulation of the OA knee following treatment with four consecutive doses (at 8 hour intervals) on giving sustained released paracetamol treatment or placebo will be compared. The fMRI and pain assessments will occur approximately 2-5 hours after taking the final dose.

DETAILED DESCRIPTION:
The objective of this study is to investigate if functional magnetic response imaging (fMRI) can detect the effects of a known pain medicine at over-the-counter doses in people with osteoarthritis (OA) of the knee. The fMRI is a harmless and painless technique that is used in the current study to collect images of brain activity to see if is changed when feeling pain. In this study, BOLD response to mechanical stimulation via pressure stimuli applied to the tibio-femoral joint and patello-femoral in participants with knee OA following four treatment doses of any of three treatment will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteoarthritis of at least one knee for 3 months
* Male or female at least 45 years of age
* Score a minimum of 4 out of 10 on the numerical pain rating and a maximum of 8 at screening

Exclusion Criteria:

* If female, is pregnant, lactating, or breast feeding
* Has secondary cause of knee arthritis
* Lower extremity surgery in the last 6 months
* Prior injury in the last twelve months to the index knee
* Used any analgesics (NSAIDs, COX2 inhibitor, etc) within 5 half lives of study start
* Recently used oral or injected glucocorticoids

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-09-01; Primary Completion 2011-08-01 (Actual); Study Completion 2011-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Hospital Del Mar, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at a single centre in Spain.
Pre-assignment Details: Out of 33 screened participants, 31 were randomized, while 2 participants were considered as screen failures
Groups:
- Sequence 1: Participants took part in 3 study sessions. Session 1-participant took two 665 mg sustained release paracetamol formulations orally with 150 ml water. Four consecutive doses were administered every 8h, with the first dose (0h) and last dose (24h) under supervision at clinic and the second dose (8h) and third dose (16h) self-administered. Session 2-no treatment was given. Session 3-participant took two caplets of matched placebo orally with 150 ml water. Four consecutive doses were administered every 8h, with the first dose (0h) and last dose (24h) under supervision at clinic and the second dose (8h) and third dose (16h) self-administered. A 5-14 day washout was given after session 1 and session 2. A 7-14 day follow-up was done after session 3.
- Sequence 2: Participants took part in 3 study sessions. Session 1-participants took two caplets of matched placebo orally with 150 ml water. Four consecutive doses were administered every 8h, with the first dose (0h) and last dose (24h) under supervision at clinic and the second dose (8h) and third dose (16h) self-administered. Session 2-no treatment was given. Session 3-participant took two 665 mg sustained release paracetamol formulations orally with 150 ml water. Four consecutive doses were administered every 8h, with the first dose (0h) and last dose (24h) under supervision at clinic and the second dose (8h) and third dose (16h) self-administered. A 5-14 day washout was given after session 1 and session 2. A 7-14 day follow-up was done after session 3.
- Sequence 3: Participants took part in 3 study sessions. Session 1-no treatment was given. Session 2-participant took two 665 mg sustained release paracetamol formulations orally with 150 ml water. Four consecutive doses were administered every 8h, with the first dose (0h) and last dose (24h) under supervision at clinic and the second dose (8h) and third dose (16h) self-administered. Session 3-participants took two caplets of matched placebo orally with 150 ml water. Four consecutive doses were administered every 8h, with the first dose (0h) and last dose (24h) under supervision at clinic and the second dose (8h) and third dose (16h) self-administered.A 5-14 day washout was given after session 1 and session 2. A 7-14 day follow-up was done after session 3.
- Sequence 4: Participants took part in 3 study sessions. Session 1-no treatment was given. Session 2-participants took two caplets of matched placebo orally with 150 ml water. Four consecutive doses were administered every 8h, with the first dose (0h) and last dose (24h) under supervision at clinic and the second dose (8h) and third dose (16h) self-administered. Session 3-participant took two 665 mg sustained release paracetamol formulations orally with 150 ml water. Four consecutive doses were administered every 8h, with the first dose (0h) and last dose (24h) under supervision at clinic and the second dose (8h) and third dose (16h) self-administered. A 5-14 day washout was given after session 1 and session 2. A 7-14 day follow-up was done after session 3.
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 8 | 7 | 8
Completed | 8 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Wash-out Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 8 | 7 | 7
Completed | 8 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 8 | 7 | 7
Completed | 7 | 8 | 7 | 7
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Wash-out Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 8 | 7 | 7
Completed | 7 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 8 | 7 | 7
Completed | 7 | 6 | 7 | 7
Not Completed | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Participants for Baseline Measurement: All randomized participants except one were evaluated for baseline measures. One participant had misallocated treatments that could not be determined. Therefore, this participant was excluded from all populations including safety.
Arm/Group | Total Participants for Baseline Measurement
Number analyzed (Participants) | 30
Age, Customized [Mean (Standard Deviation); unit: Years]
  Years | 68.5 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygen Level-Dependent (BOLD) Response in the Tibio-femoral Joint of Knee Osteoarthritis (OA): [BOLD (T-f)]
Description: BOLD response to painful pressure stimuli was evaluated using fMRI. Voxel-wise BOLD scores were reported on a Z-scale (Gaussian,mean=0,SD=1); range -3 (worst score, lowest connectivity) to +3 (best score, highest connectivity). The software derived scores compared the intensity reading in the region to a template, specifically the Montreal Neurological Institute (MNI) Echo-Planar Image (EPI) template. The template provides, for each region, expected (mean/median) intensity for that region, along with expected variation. The BOLD score on the Z-scale represents how far the actual measured intensity is from the expected in the template. A score of 0 would correspond to the mean/median, a score of 1.65 would represent the 90-percentile, -1.65 the 10-percentile, and so on, according to a standard normal distribution.
Time Frame: Baseline to 2-5 hours post last dose administration
Population: Intention-to-treat (ITT) population: all participants per period who received at least one treatment and had at least one post-baseline efficacy assessment. Missing data was not imputed.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Paracetamol 665 mg: Participants took two 665 mg Paracetamol sustained release caplets orally with 150 mL of water.
- Placebo: Participants took two placebo caplets to match Paracetamol sustained release caplets orally with 150 mL of water.
- No Treatment: No treatment was given to participants.
Arm/Group | Paracetamol 665 mg | Placebo | No Treatment
Number analyzed (Participants) | 20 | 23 | 23
Z-score | NA (NA) — BOLD value had no detectable signal for Paracetamol 665 mg group. | NA (NA) — BOLD value had no detectable signal for Placebo group. | NA (NA) — BOLD value had no detectable signal for No Treatment group.

2. Secondary Outcome: BOLD Response in the Patello-femoral Joint of Knee Osteoarthritis: [BOLD (P-f)]
Description: as for outcome 1
Time Frame: Baseline to 2-5 hours post last dose administration
Population: ITT population: all participants per period who received at least one treatment and had at least one post-baseline efficacy assessment. Missing data was not imputed.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Paracetamol 665 mg | Placebo | No Treatment
Number analyzed (Participants) | 20 | 23 | 23
Z-score
  BOLD - Sensory Cortex (a) | 0.16 (0.36) | NA (NA) — BOLD - Sensory Cortex (a) value had no detectable signal for Placebo Group. | 0.48 (0.48)
  BOLD - Supramarginal Gyrus | 0.46 (0.48) | NA (NA) — BOLD - Supramarginal Gyrus value had no detectable signal for Placebo Group. | 0.76 (0.49)
  BOLD - Thalamus | 0.48 (1.34) | -0.68 (1.74) | NA (NA) — BOLD - Thalamus value had no detectable signal for No treatment group.
  BOLD - Subgenu Prefrontal | NA (NA) — BOLD - Subgenu Prefrontal value had no detectable signal for Paracetamol 665 mg group. | -0.27 (0.41) | 0.19 (0.37)
  BOLD - Frontal Cortex | NA (NA) — BOLD - Frontal Cortex value had no detectable signal for Paracetamol 665 mg group. | -0.04 (0.31) | 0.26 (0.42)
  BOLD - Insula | NA (NA) — BOLD - Insula value had no detectable signal for Paracetamol 665 mg group. | 0.12 (0.51) | 0.62 (0.62)
  BOLD - Sensory Cortex (b) | NA (NA) — BOLD - Sensory Cortex (b) value had no detectable signal for Paracetamol 665 mg group. | -0.11 (0.60) | 0.44 (0.48)

3. Secondary Outcome: Subjective Numerical Rating Scale (NRS) Response for Treatment Effect on OA Knee Before Stimulation: [NRS (TRT)]
Description: Subjective NRS response for each participant was calculated as difference of pre-treatment NRS pain assessment before stimulus and post-treatment NRS pain assessment before stimulus. NRS responses was based on an 11 scale rating (0-10), with 0 corresponding to "No Pain" and 10 corresponding to "Extreme Pain or Pain as bad as you can imagine".
Time Frame: Baseline and post-dose before stimulus
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Paracetamol 665 Milligram (mg): Participants took two 665 mg Paracetamol sustained release caplets orally with 150mL of water.
Arm/Group | Paracetamol 665 Milligram (mg) | Placebo | No Treatment
Number analyzed (Participants) | 20 | 23 | 23
Score on a Scale | 0.95 (1.67) | -0.52 (1.53) | 0.48 (1.83)

4. Secondary Outcome: Subjective NRS Response for Treatment Effect on Tibio-femoral Stimulation Prior the fMRI Scan: [NRS (T-f Pre-scan)]
Description: Subjective NRS response was calculated for each participant as difference of pre-treatment pain assessment after stimulus and post-treatment pre-scan pain assessment after stimulus on tibio-femoral joint. NRS responses was based on an 11 scale rating (0-10), with 0 corresponding to "No Pain" and 10 corresponding to "Extreme Pain or Pain as bad as you can imagine".
Time Frame: Baseline and post-dose pre-scan after stimulus
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Paracetamol 665 mg | Placebo | No Treatment
Number analyzed (Participants) | 20 | 23 | 23
Score on a Scale | 0.55 (0.89) | 0.17 (1.07) | 0.00 (0.74)

5. Secondary Outcome: Subjective NRS Response for Treatment Effect on Patello-femoral Stimulation Prior the fMRI Scan: [NRS (P-f Pre-scan)]
Description: Subjective NRS response was calculated for each participant as difference of pre-treatment pain assessment after stimulus and post-treatment pre-scan pain assessment after stimulus on patello-femoral. NRS responses was based on an 11 scale rating (0-10), with 0 corresponding to "No Pain" and 10 corresponding to "Extreme Pain or Pain as bad as you can imagine".
Time Frame: Baseline and post-dose pre-scan after stimulus
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Paracetamol 665 mg | Placebo | No Treatment
Number analyzed (Participants) | 20 | 23 | 23
Score on a Scale | 0.60 (1.23) | 0.43 (0.95) | 0.00 (0.91)

6. Secondary Outcome: Subjective NRS Response for Treatment Effect on Tibio-femoral Stimulation After the fMRI Scan: [NRS (T-f Post-scan)]
Description: Subjective NRS response for treatment effect on tibio-femoral stimulus after the fMRI scan was calculated for each participant as difference of pre-treatment pain assessment after stimulus and post-treatment post-scan pain assessment after stimulus on tibio-femoral. NRS responses was based on an 11 scale rating (0-10), with 0 corresponding to "No Pain" and 10 corresponding to "Extreme Pain or Pain as bad as you can imagine".
Time Frame: Baseline and post-dose post-scan after stimulus
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Paracetamol 665 mg | Placebo | No Treatment
Number analyzed (Participants) | 20 | 23 | 23
Score on a Scale | 0.15 (1.18) | 0.09 (1.38) | -0.13 (1.10)

7. Secondary Outcome: Subjective NRS Response for Treatment Effect on Patello-femoral Stimulation After the fMRI Scan: [NRS (P-f Post-scan)]
Description: Subjective NRS response for each participant for treatment effect on tibio-femoral stimulus after the fMRI scan was calculated as difference of pre-treatment pain assessment after stimulus and post-treatment post-scan pain assessment after stimulus on patello-femoral. NRS responses was based on an 11 scale rating (0-10), with 0 corresponding to "No Pain" and 10 corresponding to "Extreme Pain or Pain as bad as you can imagine".
Time Frame: Baseline and post-dose post-scan after stimulus
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Paracetamol 665 mg | Placebo | No Treatment
Number analyzed (Participants) | 20 | 23 | 23
Score on a Scale | 0.30 (1.66) | -0.48 (1.62) | -0.39 (1.92)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of start of the investigational product, and until 5 days following last administration of the investigational product.
Arm/Group | Paracetamol 665 mg | Placebo | No Treatment
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 3/29 | 3/28 | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paracetamol 665 mg (N=29) | Placebo (N=28) | No Treatment (N=30)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Claustrophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.